CLINICAL TRIAL: NCT01471522
Title: International Study of Comparative Health Effectiveness With Medical and Invasive Approaches (ISCHEMIA)
Acronym: ISCHEMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York University (Other); Stanford University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Albany Stratton VA Medical Center (U.S. Federal Agency); Cedars-Sinai Medical Center (Other); Columbia University (Other); Duke University (Other); East Carolina University (Other); Emory University (Other); Harvard University (Other); Massachusetts General Hospital (Other); Montreal Heart Institute (Other); University of British Columbia (Other); University of Missouri, Kansas City (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-00498; 1U01HL105907 (NIH)
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia | interventions — Cardiac Catheterization; Coronary Artery Bypass; Percutaneous Coronary Intervention; Dosage Forms; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Invasive Strategy (INV) (Active Comparator): Routine invasive strategy with cardiac catheterization followed by revascularization plus optimal medical therapy.
  Interventions: Procedure: cardiac catheterization; Procedure: coronary artery bypass graft surgery; Procedure: percutaneous coronary intervention; Behavioral: Lifestyle; Drug: Medication
- Conservative Strategy (Active Comparator): Optimal medical therapy with cardiac catheterization and revascularization reserved for patients with acute coronary syndrome, ischemic heart failure, resuscitated cardiac arrest or refractory symptoms.
  Interventions: Behavioral: Lifestyle; Drug: Medication

INTERVENTIONS:
Procedure: cardiac catheterization — Narrowed blood vessels can be opened without surgery using stents or can be bypassed with surgery. To determine which is the best approach for you the doctor needs to look at your blood vessels to see where the narrowings are and how much narrowing there is. This is done by a procedure known as a cardiac catheterization.
  Other Names: cath
  Arms: Invasive Strategy (INV)
Procedure: coronary artery bypass graft surgery — Artery narrowing is bypassed during surgery with a healthy artery or vein from another part of the body. This is known as coronary artery bypass grafting, or CABG (said, "cabbage"). The surgery creates new routes around narrowed and blocked heart arteries. This allows more blood flow to the heart.
  Other Names: CABG
  Arms: Invasive Strategy (INV)
Procedure: percutaneous coronary intervention — Percutaneous coronary intervention may be done as part of the cardiac catheterization procedure. With this procedure a small, hollow, mesh tube (stent) is inserted into the narrowed part of the artery. The stent pushes the plaque against the artery wall, and opens the vessel to allow better blood flow.
  Other Names: PCI
  Arms: Invasive Strategy (INV)
Behavioral: Lifestyle — diet, physical activity, smoking cessation
  Other Names: Behavior change
Drug: Medication — antiplatelet, statin, other lipid lowering, antihypertensive, and anti-ischemic medical therapies
  Other Names: Pharmacologic Therapy

SUMMARY:
The purpose of the ISCHEMIA trial is to determine the best management strategy for higher-risk patients with stable ischemic heart disease (SIHD). This is a multicenter randomized controlled trial with 5179 randomized participants with moderate or severe ischemia on stress testing. A blinded coronary computed tomography angiogram (CCTA) was performed in most participants with eGFR ≥60 mL/min/1.73m2 to identify and exclude participants with either significant unprotected left main disease (≥50% stenosis) or those without obstructive CAD (<50% stenosis in all major coronary arteries). Of 8518 participants enrolled, those that had insufficient ischemia, ineligible anatomy demonstrated on CCTA or another exclusion criterion, did not go on to randomization. Eligible participants were then assigned at random to a routine invasive strategy (INV) with cardiac catheterization followed by revascularization, if feasible, plus optimal medical therapy (OMT) or to a conservative strategy (CON) of OMT, with cardiac catheterization and revascularization reserved for those who fail OMT.

SPECIFIC AIMS

A. Primary Aim The primary aim of the ISCHEMIA trial is to determine whether an initial invasive strategy of cardiac catheterization followed by optimal revascularization, if feasible, in addition to OMT, will reduce the primary composite endpoint of cardiovascular death, nonfatal myocardial infarction, resuscitated cardiac arrest, or hospitalization for unstable angina or heart failure in participants with SIHD and moderate or severe ischemia over an average follow-up of approximately 3.5 years compared with an initial conservative strategy of OMT alone with catheterization reserved for failure of OMT.

B. Secondary Aims Secondary aims are to determine whether an initial invasive strategy compared to a conservative strategy will improve: 1) the composite of CV death or MI; 2) angina symptoms and quality of life, as assessed by the Seattle Angina Questionnaire; 3) all-cause mortality; 4) net clinical benefit assessed by including stroke in the primary and secondary composite endpoints; and 5) individual components of the composite endpoints.

Condition: Coronary Disease Procedure: Coronary CT Angiogram Procedure: Cardiac catheterization Phase: Phase III per NIH

Condition: Cardiovascular Diseases Procedure: Angioplasty, Transluminal, Percutaneous Coronary, other catheter-based interventions Phase: Phase III per NIH

Condition: Heart Diseases Procedure: Coronary Artery Bypass Surgery Phase: Phase III per NIH

DETAILED DESCRIPTION:
BACKGROUND:

Evidence supporting a routine invasive practice paradigm for patients with SIHD is outdated. In strategy trials conducted in the 1970s, coronary artery bypass grafting (CABG) improved survival as compared with no CABG in SIHD patients with high-risk anatomic features. The relevance of these studies today is speculative because contemporary secondary prevention-aspirin, beta-blockers, statins, ACE inhibitors, and lifestyle interventions-were used minimally if at all. Subsequent trials have compared percutaneous coronary intervention (PCI) with medical therapy, as PCI has replaced CABG as the dominant method of revascularization for SIHD. To date, PCI has not been shown to reduce death or myocardial infarction (MI) compared with medical therapy in SIHD patients.

COURAGE and BARI 2D, the two largest trials comparing coronary revascularization vs. medical therapy in SIHD patients, found that among patients selected on the basis of coronary anatomy after cardiac catheterization, an initial management strategy of coronary revascularization (PCI, PCI or CABG, respectively) did not reduce the primary endpoints of death or MI (COURAGE), or death (BARI 2D) compared with OMT alone. These data suggest, but do not prove, that routine cardiac catheterization--which often leads to ad hoc PCI through the diagnostic-therapeutic cascade--may not be required in SIHD patients. However, most patients enrolled in COURAGE and BARI 2D who had ischemia severity documented at baseline had only mild or moderate ischemia, leaving open the question of the appropriate role of cardiac catheterization and revascularization among higher-risk patients with more severe ischemia. Observational data suggest that revascularization of patients with moderate-to-severe ischemia is associated with a lower mortality than medical therapy alone, but such data cannot establish a cause and effect relationship. In clinical practice only about half such patients are referred for cardiac catheterization, indicating equipoise. Furthermore, analysis of outcomes for 468 COURAGE patients with moderate-to-severe ischemia at baseline did not reveal a benefit from PCI. This issue cannot be resolved using available data because all prior SIHD strategy trials enrolled patients after cardiac catheterization, introducing undefined selection biases (e.g., highest risk patients not enrolled) and making translation of study results problematic for clinicians managing patients who have not yet had cardiac catheterization.

A clinical trial in SIHD patients uniformly at higher risk (which could not have been performed before COURAGE and BARI 2D results were available) is needed to inform optimal management for such patients.

DESIGN NARRATIVE, INCLUDING MODIFICATIONS DURING THE TRIAL

Primary Endpoint

A composite of CV death, MI, resuscitated cardiac arrest, or hospitalization for unstable angina or heart failure was proposed as the primary endpoint in the application that was funded by NLHBI, with a secondary endpoint of CV death or MI. Study protocol version 1.0 was finalized on January 18, 2012 after review and approval by the protocol review committee (DSMB) with the primary endpoint specified as the composite of CV death or MI. Regarding the final status of the primary endpoint, the protocol stated:

"To ensure that the primary analysis is well-powered and useful, a prospective plan to allow extending follow-up and/or changing the primary endpoint based on aggregate event rate data will be established prior to the first review of unblinded trial data. At a designated time during the trial, an analysis will be conducted to estimate the overall aggregate primary endpoint event rate and project the final number of observed events. If the estimated unconditional power (i.e. based on aggregate event rate data; not by treatment group) is less than the originally targeted 90%, then one or more of the following options will be considered:

1. Extend follow-up to allow more events to accrue.
2. Change the primary endpoint to one that occurs more frequently. The current primary endpoint would become a secondary endpoint. The proposed new primary endpoint would be the composite of CV death, MI, resuscitated cardiac arrest, or hospitalization for unstable angina or heart failure.
3. Follow the recommendation of an independent advisory panel. An independent advisory panel, separate from the DSMB, will be convened for the purpose of reviewing unconditional power estimates and making a recommendation to the NHLBI Director. Members of this panel will not have access to unblinded data by treatment group or other data that may bias their recommendation." All 5 event types were adjudicated throughout the trial. Study protocol v2.0 (January 2014) allowed ischemia eligibility by non-imaging exercise stress test if more stringent (≥70% stenosis) CCTA criteria were met. The 2016 protocol addendum describes the NHLBI-approved reduction in sample size and extension of recruitment and follow-up due to slower than projected recruitment.

The pre-specified first analysis for monitoring and projecting the final aggregate number of primary endpoint events was conducted in 2015. In 2016, the projected need to increase the power by extending follow-up and elevating the 5-component secondary endpoint to become primary was discussed at Steering Committee and Investigator meetings and communicated by email.

An Independent Advisory Panel convened by NHLBI met in May 2017, and in June 2017 NHLBI approved the Independent Advisory Panel's recommendation to elevate the 5-component secondary endpoint to become primary and retain the 2-component composite as a key secondary endpoint. The panel also recommended extension of follow-up. This was communicated to the Steering Committee and Investigators at August and November 2017 meetings and by email. The last visit date was June 30, 2019.

A statistical plan developed for the Independent Advisory Panel process in 2012 specified that a decision about changing the primary endpoint would be targeted to occur before 75% of the final number of primary endpoint events had accrued. Although the final number of primary endpoint events was unknown during the course of the trial, estimates performed at the time of the Advisory Panel meeting suggested that the ratio of accrued endpoint events to final endpoint events was below 50%. See Maron DJ et al. Am Heart J. 2018 201:124-135. PMC6005768 for additional details about modifications to the trial while it was being conducted.

Analysis of Patients' Health Status as a Key Secondary Endpoint

A key secondary objective of the ISCHEMIA trial is to compare the quality of life outcomes-patients' symptoms, functioning and well-being-between those assigned to an invasive strategy as compared with a conservative strategy. In the protocol, angina frequency and disease-specific quality of life measured by the Seattle Angina Questionnaire (SAQ) Angina Frequency and Quality of Life scales, respectively, are described as the tools that will be used to make this comparative assessment. Recent work has indicated that it is possible to combine the information from the individual domain scores in the SAQ into a new Summary Score that captures the information from the SAQ Angina Frequency, Physical Limitation and Quality of Life scales into a single overall score. The advantages of using a summary score as the primary measure of QOL effects of a therapy are a single primary endpoint comparison rather than two or three (eliminating concerns some may have about multiple comparisons) and a more intuitive holistic (patient-centric) interpretation of the effectiveness results. With these advantages in mind, the ISCHEMIA leadership has agreed that the SAQ Summary Score will be designated as the primary way this outcome for this key secondary endpoint of the ISCHEMIA trial will be analyzed and interpreted, with the individual SAQ scores being used in a secondary, explanatory and descriptive role.

PARTICIPATING COUNTRIES:

North America:

Canada; Mexico; USA

South America:

Argentina; Brazil; Peru

Asia:

China; India; Japan; Malaysia; Singapore; Taiwan; Thailand; Russian Federation

Pacifica:

Australia; New Zealand

Europe:

Austria; Belgium; France; Germany; Hungary; Italy; Lithuania; Macedonia; Netherlands; Poland; Portugal; Romania; Serbia; Spain; Sweden; Switzerland; UK

Middle East:

Egypt; Israel; Saudi Arabia

Africa:

South Africa

ELIGIBILITY:
Inclusion Criteria:

* At least moderate ischemia on a qualifying stress test
* Participant is willing to comply with all aspects of the protocol, including adherence to the assigned strategy, medical therapy and follow-up visits
* Participant is willing to give written informed consent
* Age ≥ 21 years

Exclusion Criteria:

* LVEF < 35%
* History of unprotected left main stenosis >50% on prior coronary computed tomography angiography (CCTA) or prior cardiac catheterization (if available)
* Finding of "no obstructive CAD" (<50% stenosis in all major epicardial vessels) on prior CCTA or prior catheterization, performed within 12 months
* Coronary anatomy unsuitable for either PCI or CABG
* Unacceptable level of angina despite maximal medical therapy
* Very dissatisfied with medical management of angina
* History of noncompliance with medical therapy
* Acute coronary syndrome within the previous 2 months
* PCI within the previous 12 months
* Stroke within the previous 6 months or spontaneous intracranial hemorrhage at any time
* History of ventricular tachycardia requiring therapy for termination, or symptomatic sustained ventricular tachycardia not due to a transient reversible cause
* NYHA class III-IV heart failure at entry or hospitalization for exacerbation of chronic heart failure within the previous 6 months
* Non-ischemic dilated or hypertrophic cardiomyopathy
* End stage renal disease on dialysis or estimated glomerular filtration rate (eGFR) <30mL/min (not an exclusion criterion for CKD ancillary trial, see CKD ancillary trial, Section 18)
* Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial
* Allergy to radiographic contrast that cannot be adequately pre-medicated, or any prior anaphylaxis to radiographic contrast
* Planned major surgery necessitating interruption of dual antiplatelet therapy (note that patients may be eligible after planned surgery)
* Life expectancy less than the duration of the trial due to non-cardiovascular comorbidity
* Pregnancy (known to be pregnant; to be confirmed before CCTA and/or randomization, if applicable)
* Patient who, in the judgment of the patient's physician, is likely to have significant unprotected left main stenosis (Those who are able to undergo CCTA will have visual assessment of the left main coronary artery by the CCTA core lab)
* Enrolled in a competing trial that involves a non-approved cardiac drug or device
* Inability to comply with the protocol
* Exceeds the weight or size limit for CCTA or cardiac catheterization at the site
* Canadian Cardiovascular Society Class III angina of recent onset, OR angina of any class with a rapidly progressive or accelerating pattern
* Canadian Cardiovascular Society Class IV angina, including unprovoked rest angina
* High risk of bleeding which would contraindicate the use of dual antiplatelet therapy
* Cardiac transplant recipient
* Prior CABG, unless CABG was performed more than 12 months ago, and coronary anatomy has been demonstrated to be suitable for PCI or repeat CABG to accomplish complete revascularization of ischemic areas (CCC approval required)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5179 (Actual)
Dates: Start 2012-07; Primary Completion 2019-06-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Hochman, MD, Study Chair — New York University; David J Maron, MD, Principal Investigator — Stanford University
Locations (320):
- United States (109):
  - UAB Vascular Biology and Hypertension Program, Birmingham, Alabama
  - Yuma Regional Medical Center, Yuma, Arizona
  - Cedars Sinai Medical Center, Beverly Hills, California
  - UCSF - Fresno Community Regional Medical Center, Fresno, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - VA Palo Alto HealthCare System, Palo Alto, California
  - Kaiser Permanente San Jose, San Jose, California
  - Coastal Heart Medical Group, Santa Ana, California
  - Stanford University School of Medicine, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - South Denver Cardiology Associates, P.C., Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Daytona Heart Group, Daytona Beach, Florida
  - Malcom Randall VAMC, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Advanced Heart Care Group, Fairview Heights, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University/Krannert Institute of Cardiology, Indianapolis, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Lexington VA Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Cardiovascular Specialists of Southwest Louisiana, Lake Charles, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham & Women's Hospital, Harvard Medical School, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - VA Boston Healthcare System, West Roxbury, Massachusetts
  - Saint Vincent Hospital at Worcester Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Providence - Providence Park Hospital, Southfield, Michigan
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Minneapolis VAMC, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - HealthEast Saint Joseph's Hospital, Saint Paul, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Hackensack University Medical Center, Saddle Brook, New Jersey
  - Albany Medical Center Hospital, Albany, New York
  - Samuel Stratton VA Medical Center of Albany NY, Albany, New York
  - Capital Cardiology Associates, Albany, New York
  - NYU-HHC Kings County Hospital Center, Brooklyn, New York
  - New York -Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - NYU-HHC Woodhull Hospital, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - NYP Medical Medical Group Hudson Valley Cardiology, Cortlandt Manor, New York
  - New York University - Langone Cardiovascular Associates, Flushing, New York
  - Mid Valley Cardiology, Kingston, New York
  - Northwell Health - Manhasset, Manhasset, New York
  - NYU Winthrop, Mineola, New York
  - VA New York Harbor Health Care System, New York, New York
  - Beth Israel Medical Center, New York, New York
  - NYU Langone Medical Center-Bellevue Hospital, New York, New York
  - NYU New York Medical Associates, New York, New York
  - Mount Sinai Saint Luke's Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Cardiology Associates of Schenectady P.C., Schenectady, New York
  - NYU-HHC Lincoln Medical and Mental Health Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Louis Stokes Cleveland Veterans Affairs Medical Center, Cleveland, Ohio
  - Ohio Health Grant Medical Center, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Saint Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Holy Spirit Hospital Cardiovascular Institute, Camp Hill, Pennsylvania
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Conemaugh Valley Memorial Hospital, Johnstown, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - V.A. North Texas Health Care System, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Heart & Vascular Associates, Houston, Texas
  - Baylor Research Institute at Legacy Heart Center, Plano, Texas
  - The Heart Hospital Baylor, Plano, Texas
  - Audie Murphy V.A., San Antonio, Texas
  - Medicus Alliance Clinical Research Org., Inc., Sugar Land, Texas
  - Wichita Falls Heart Clinic, Wichita Falls, Texas
  - Salt Lake City VA Medical Center, Salt Lake City, Utah
  - VAMC-White River Junction, White River Junction, Vermont
  - Cardiovascular Associates, Ltd., Chesapeake, Virginia
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Winchester Cardiology and Vascular Medicine, PC, Winchester, Virginia
  - University of Washington Medical Center, Bellevue, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
- Argentina (6):
  - Hospital Italiano Regional del Sur Bahia Blanca, Bahía Blanca, Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Medico DAMIC, Córdoba, CBA
  - Clinica Del Prado, Córdoba
  - Clinica Romagosa and Clinica De La Familia, Córdoba
  - Clínica Privada Vélez Sarsfield, Córdoba
- Australia (4):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - LKH Graz West Austria, Graz, Stmk
  - Medical University of Vienna, Department of Cardiology, Vienna, Vienna
  - Wilhelminen Hospital Vienna, Vienna, Vienna
- University Hospital Leuven, Leuven, Brabant, Belgium
- Brazil (17):
  - Fundacao Bahiana de Cardilogia, Salvador, Estado de Bahia
  - Hospital Lifecenter, Belo Horizonte, Minas Gerais
  - Hospital Maternidade e Pronto Socorro Santa Lucia, Poços de Caldas, Minas Gerais
  - Quanta Diagnostico & Terapia, Curitiba, Paraná
  - Hospital Cardiologico Costantini, Curitiba, Paraná
  - Hospital Pró-Cardíaco, Botafogo, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sol, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto Dante Pazzanese de Cardiologia, Ibirapuera, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Hospital TotalCor, São Paulo, São Paulo
  - Hospital da Bahia, Salvador
  - Unifesp - Hospital Sao Paulo, São Paulo
  - Heart Institute (InCor) University of São Paulo, São Paulo
  - Hospital Celso Pierro, São Paulo
- Canada (19):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - West Lincoln Memorial Hospital, Grimsby, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Dixie Medical Group, Mississauga, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Saint Catharines General Hospital, St. Catharines, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Northwest GTA Cardiovascular and Heart Rhythm Program, Vaughan, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux du Montréal, Montreal, Quebec
  - CISSSL - Hopital Pierre-Le Gardeur, Terrebonne, Quebec
  - Centre Hospitalier de Regional Trois-Rivieres, Trois-Rivières, Quebec
  - University of Ottawa Heart Institute, Ottawa
- China (20):
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Chaoyang
  - Liangxiang Hospital, Beijing Fangshan District, Beijing, Fangshan
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Medical College, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Tongji Medical College, Huazhong Science and Tech University, Wuhan, Hubei
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Qingdao Fuwai Hospital, Qingdao, Shandong
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Xian, Shanxi
  - TEDA International Cardiovascular Hospital, Tianjing, Tianjing
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Cairo University, Cairo, Egypt
- France (7):
  - C.H. Louis Pasteur, Châtres, Centre-Val de Loire
  - Grenoble University Hospital, Grenoble, Isere
  - Centre Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Ambroise Pare Hospital, Boulogne-Billancourt, Île-de-France Region
  - Antoine-Beclere Hospital, Clamart, Île-de-France Region
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes, Île-de-France Region
  - Bichat Hospital, Paris, Île-de-France Region
- Germany (4):
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Universitatsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Praxisklinik Herz Und Gefaesse, Dresden, Saxony
  - University Hospital Jena, Jena, Thuringia
- Hungary (5):
  - University of Szeged, Szeged, Szeged Megyei Varos
  - Eszszk- Szent Istvan Hospital, Budapest
  - Military Hospital, Budapest, Budapest
  - Heart and Vascular Center, Semmelweis University, Budapest
  - George Gottsegen National Institute of Cardiology, Budapest
- India (19):
  - Gurunanak CARE Hospital, Hyderabad, Andhra Pradesh
  - CARE Hospital, Hyderabad, Andhra Pradesh
  - Sri Jayadeva Institute of Cardiovascular Sciences and Research, Bangalore, Karnataka
  - Government Medical College, Calicut, Kerala
  - MOSC Medical College Hospital, Kolenchery, Kolenchery, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Trivandrum, Kerala
  - Ruby Hall Clinic,Grant Medical Foundation, Pune, Maharashtra
  - KEM Hospital Pune, Pune, Maharashtra
  - Dr Ram Manohar Lohia Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Escort Heart Institute, New Delhi, National Capital Territory of Delhi
  - Batra Hospital and Medical Research Centre (BHMRC), New Delhi, National Capital Territory of Delhi
  - Fortis Healthcare Fl.t Lt. Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi
  - Hero DMC Heart Institute, Dayanand Medical College and Hospital, Ludhiana, Punjab
  - Apollo Research and Innovation, Chennai, Tamil Nadu
  - Jawaharlal Institute of Postgraduate Medical Education & Research (JIPMER), Pondicherry, Tamil Nadu
  - CARE Nampally, Hyderabad, Telangana
  - Apollo Research & Innovations, Hyderabad, Telangana
  - King George's Medical University, Department of Cardiology, Lucknow, Uttar Pradesh
  - All India Institute of Medical Sciences, New Delhi
- Israel (2):
  - Rambam Medical Center, Haifa
  - Assuta Medical Centers, Tel Aviv
- Italy (13):
  - AORN Dei Colli "V. Monaldi" UOC Cardiologia Università della Campania "L.Vanvitelli", Napoli, Campania
  - Ospedale "G.B. Morgagni - L. Pierantoni" Forli (AUSL della Romagna), Forlì, Emilia-Romagna
  - IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo, FG
  - Policlinico di Monza, Monza MB, Monza, MB
  - Humanitas Research Hospital, Rozzano (MI), Rozzano, Milano
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, Piedmont
  - Cardiology and CCU - Ospedali Riuniti Ancona, Ancona, The Marches
  - UO Cardiologia Ospedale SS Cosma e Damiano, Pescia, Tuscany
  - Azienda Servizi Sanitaria n.3 Alto Friuli-Collinare-Medio Friuli, Tolmezzo, Udine
  - University of Padua- Cardiology Clinic, Padua, Veneto
  - Ospedale Regionale Umberto Parini, Aosta
  - Clinica Mediterranea, Naples
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (3):
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Saitama Medical University, Hidaka, Saitama
  - Keio University Hospital, Shinjuku-Ku, Tokyo
- Vilnius University Hospital Santariskes Clinic, Vilnius, Lithuania
- Institut Jantung Negara, Kuala Lumpur, Kuala Lumpur, Malaysia
- Mexico (2):
  - Instituto Mexicano del Seguro Social, Benito Juárez, Mexico City
  - Instituto Nacional de Cardiología "Ignacio Chávez", Mexico City, Mexico City
- Netherlands (3):
  - Cardio Research Hartcentrum OLVG, Amsterdam, North Holland
  - Radboudumc, Nijmegen
  - Isala Klinieken, Zwolle
- New Zealand (2):
  - Waikato Hospital, Hamilton, Waikato Region
  - Auckland City Hospital, Auckland
- University Clinic of Cardiology, Skopje, Republic of Macedo, North Macedonia
- Instituto Neuro Cardiovascular De Las Americas, Miraflores, Lima region, Peru
- Poland (12):
  - T.Marciniak Hospital, Wroclaw, Dolny Śląsk
  - Department of Coronary Disease, John Paul II Hospital, Jagiellonian University Medical College, Krakow, Maopolskie
  - Department of Internal Medicine and Cardiology, Infant Jesus Teaching Hospital, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Coronary and Structural Heart Diseases Department, Institute of Cardiology, Warsaw, Masovian Voivodeship
  - Department of Interventional Cardiology & Angiology, Institute of Cardiology, Warsaw, Masovian Voivodeship
  - Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Institute of Cardiology, Warsaw, Warsaw, Mazovian
  - University Hospital in Bialystok, Bialystok, Podlaskie Voivodeship
  - Medical University of Silesia, School of Medicine with the Division of Dentistry, Department of Cardiology, Congenital Heart Diseases and Electrotherapy, Silesian Center for Heart Diseases, Zabrze, Silesian Voivodeship
  - Szpital Kliniczny Przemienienia Pańskiego, Poznan
  - Military Hospital / Medical University, Wroclaw
  - Cardiology Clinic, Medical University in Lodz, Lodz, Łódź Voivodeship
- Portugal (3):
  - Hospital de Santa Marta, Lisbon
  - Santa Maria University Hospital, Cardiology Department, CHLN, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Vila Nova de Gaia
- Romania (2):
  - Emergency County Hospital Baia Mare, Baia Mare
  - Emergency Institute of Cardiovascular Diseases ''Prof. Dr. C. C. Iliescu'', Bucharest
- Russia (4):
  - National Medical Research Center for Cardiovascuar Surgery, Moscow, Gorod Moskva
  - E.Meshalkin National Medical Research Center of the Ministry of Health of the Russian Federation, Novosibirsk, Novosibirsk Oblast
  - Federal Almazov North-West Medical Research Centre, Saint Petersburg
  - North-Western State Medical University, Saint Petersburg
- King AbdulAziz Cardiac Center, Riyadh, Central Province, Saudi Arabia
- Serbia (7):
  - Institute of Cardiovascular Diseases Vojvodina, Sremska Kamenica, Serbia and Faculty of Medicine, University of Novi Sad, Kamenitz, Vojvodina
  - Clinical Center of Serbia, Belgrade
  - Faculty of Medicine, University of Belgrade; Cardiology Clinic, Clinical Center of Serbia, Belgrade
  - University Clinical Hospital Zvezdara, Belgrade
  - University Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinic for Cardiovascular Diseases, Clinical Center Nis, Niš
- Singapore (3):
  - National University Heart Center Singapore, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- Groote Schuur Hospital / University of Cape Town, Cape Town, Western Cape, South Africa
- Spain (9):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, La Coruna
  - Complexo Hospitalario Universitario A Coruña (CHUAC) Sergas, Department of Cardiology. INIBIC A Coruña. CIBER-CV. Universidad de A Coruña, Spain, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital De Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital La Paz. IdiPaz, Madrid
  - HUVA, Hospital Clínico Universitario Virgen De La Arrixaca, Murcia
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Karolinska Institutet at Danderyd Hospital, Stockholm
  - Uppsala University, Uppsala
- Cardiocentro, Lugano, Canton Ticino, Switzerland
- Mackay Memorial Hospital, Taipei, Taiwan
- Thailand (2):
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Meung
  - Ramathibodi Hospital, Bangkok
- United Kingdom (28):
  - Belfast Trust, Belfast, Antrim
  - Bedford Hospital NHS Trust, Bedford, Bedfordshire
  - Luton and Dunstable University Hospital NHS FT, Luton, Berdfordshire
  - Papworth Hospital, Cambridge, Cambridgeshire
  - Peterborough City Hospital, Peterborough, Cambs
  - The James Cook University Hospital, Middlesbrough, Middlesbrough, Cleveland
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Dorset County Hospital, Dorchester, Dorset
  - The University of Hull/Castle Hill Hospital, Cottingham, East Yorkshire
  - Broomfield Hospital, Chelmsford, Essex
  - Southend University Hospital, Westcliff-on-Sea, Essex
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - Blackpool Teaching Hospitals, Blackpool, Lancashire
  - The Pennine Acute Hospitals NHS Trust, Oldham, Lancashire
  - Northwick Park Hospital Harrow/ Royal Brompton Hospital London, Harrow, Middlesex
  - South Eastern Health and Social Care, Belfast, Northern Ireland
  - Cardiovascular Research Unit, Craigavon Area Hospital, Craigavon, Northern Ireland
  - Nottingham University Hospitals, Nottingham, Notts
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - University of Glasgow, Clydebank, Strathclyde
  - Russells Hall Hospital, Dudley, West Midlands
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Pinderfields Hospital, Wakefield, West Yorkshire
  - University College London Hospitals NHS Foundation Trust/Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - King's College NHS Foundation Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to the NHLBI according to their guidelines within 3 years after the final patient follow-up (June 30, 2019) or 2 years after the main paper of the trial has been published, whichever comes first.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: June 2022

REFERENCES:
- [Background] Maron DJ, Stone GW, Berman DS, Mancini GB, Scott TA, Byrne DW, Harrell FE Jr, Shaw LJ, Hachamovitch R, Boden WE, Weintraub WS, Spertus JA. Is cardiac catheterization necessary before initial management of patients with stable ischemic heart disease? Results from a Web-based survey of cardiologists. Am Heart J. 2011 Dec;162(6):1034-1043.e13. doi: 10.1016/j.ahj.2011.09.001. PMID 22137077
- [Background] Phillips LM, Hachamovitch R, Berman DS, Iskandrian AE, Min JK, Picard MH, Kwong RY, Friedrich MG, Scherrer-Crosbie M, Hayes SW, Sharir T, Gosselin G, Mazzanti M, Senior R, Beanlands R, Smanio P, Goyal A, Al-Mallah M, Reynolds H, Stone GW, Maron DJ, Shaw LJ. Lessons learned from MPI and physiologic testing in randomized trials of stable ischemic heart disease: COURAGE, BARI 2D, FAME, and ISCHEMIA. J Nucl Cardiol. 2013 Dec;20(6):969-75. doi: 10.1007/s12350-013-9773-4. PMID 23963599
- [Background] ISCHEMIA Trial Research Group; Maron DJ, Hochman JS, O'Brien SM, Reynolds HR, Boden WE, Stone GW, Bangalore S, Spertus JA, Mark DB, Alexander KP, Shaw L, Berger JS, Ferguson TB Jr, Williams DO, Harrington RA, Rosenberg Y. International Study of Comparative Health Effectiveness with Medical and Invasive Approaches (ISCHEMIA) trial: Rationale and design. Am Heart J. 2018 Jul;201:124-135. doi: 10.1016/j.ahj.2018.04.011. Epub 2018 Apr 21. PMID 29778671
- [Background] Hochman JS, Reynolds HR, Bangalore S, O'Brien SM, Alexander KP, Senior R, Boden WE, Stone GW, Goodman SG, Lopes RD, Lopez-Sendon J, White HD, Maggioni AP, Shaw LJ, Min JK, Picard MH, Berman DS, Chaitman BR, Mark DB, Spertus JA, Cyr DD, Bhargava B, Ruzyllo W, Wander GS, Chernyavskiy AM, Rosenberg YD, Maron DJ; ISCHEMIA Research Group. Baseline Characteristics and Risk Profiles of Participants in the ISCHEMIA Randomized Clinical Trial. JAMA Cardiol. 2019 Mar 1;4(3):273-286. doi: 10.1001/jamacardio.2019.0014. PMID 30810700
- [Derived] Kwong RY, Heydari B, Abbasi S, Mongeon FP, Marcotte F, Friedrich M, Shaw LJ, Xu Y, Anthopolos R, Bekeredjian R, Monti L, Selvanayagam J, Lesiak M, Picard MH, Berman DS, Bangalore S, Spertus JA, Stone GW, Boden WE, Min J, Mancini GBJ, Leipsic J, Budoff M, Hague C, Hochman JS, Maron DJ, Reynolds HR; ISCHEMIA Research Group. Stress Cardiac Magnetic Resonance Ischemia Burden and Cardiovascular Events: Post-Hoc Analysis From the ISCHEMIA Trial. JACC Cardiovasc Imaging. 2025 Dec 5:S1936-878X(25)00597-2. doi: 10.1016/j.jcmg.2025.10.015. Online ahead of print. PMID 41351610
- [Derived] Ikemura N, Jones PG, Fu Z, Chan PS, Sherrod CF 4th, Arnold SV, Cohen DJ, Mark DB, Maron DJ, Hochman JS, Spertus JA; ISCHEMIA Research Group. Trajectories of Angina After Initial Invasive vs Conservative Strategy for Chronic Coronary Disease. J Am Coll Cardiol. 2025 Sep 16;86(11):782-793. doi: 10.1016/j.jacc.2025.06.044. PMID 40930615
- [Derived] Huded CP, Spertus JA, Jones PG, O'Brien SM, Mark DB, Bangalore S, Stone GW, Williams DO, White HD, Boden WE, Reynolds HR, Hochman JS, Maron DJ; ISCHEMIA Research Group. Health Status Outcomes With Percutaneous Coronary Intervention and Coronary Artery Bypass Grafting in ISCHEMIA. Circulation. 2025 Sep 23;152(12):846-858. doi: 10.1161/CIRCULATIONAHA.125.073591. Epub 2025 Sep 5. PMID 40910165
- [Derived] Shaw LJ, Phillips LM, Leipsic J, Broderick S, Mieres JH, Marwick TH, Friedrich MG, Miller T, Lopes RD, Chow B, Cerci R, Blankstein R, DiCarli M, Maron DJ, Hochman JS, Alexander KP, Stone GW, O'Brien S, Chaitman BR, Kwong RY, Picard MH, Berman DS, Reynolds HR; ISCHEMIA Research Group. Comparative Prognosis by Stress ECG and Stress Imaging: Results From the ISCHEMIA Trial. JACC Cardiovasc Imaging. 2025 Sep;18(9):943-955. doi: 10.1016/j.jcmg.2025.03.016. Epub 2025 Jul 9. PMID 40637654
- [Derived] White HD, O'Brien SM, Boden WE, Fremes SE, Bangalore S, Reynolds HR, Stone GW, Ali ZA, Parakh N, Lopez-Sendon JL, Wang Y, Chen YQ, Mark DB, Chaitman BR, Spertus JA, Maron DJ, Hochman JS; ISCHEMIA Research Group.. Use of coronary artery bypass graft surgery and percutaneous coronary intervention and associated outcomes in the ISCHEMIA trial. Am Heart J. 2025 Nov;289:78-94. doi: 10.1016/j.ahj.2025.05.009. Epub 2025 May 20. PMID 40404111
- [Derived] Lerner JB, Pleasure M, Min JK, Picard MH, Peteiro J, Senior R, Celutkiene J, Shapiro MD, Pellikka PA, de Quadros AS, Chow BJW, Tamis-Holland JE, Rodriguez F, Fleg JL, Maron DJ, Hochman JS, Reynolds HR; CIAO-ISCHEMIA Research Group. Quantitative Coronary Artery Plaque Parameters and Severity of Ischemia in Patients With INOCA. Circ Cardiovasc Imaging. 2025 Apr;18(4):e017367. doi: 10.1161/CIRCIMAGING.124.017367. Epub 2025 Mar 31. No abstract available. PMID 40163030
- [Derived] Bangalore S, Mancini GBJ, Leipsic J, Budoff MJ, Xu Y, Anthopolos R, Brilakis ES, Dwivedi A, Spertus JA, Jones PG, Cho YJ, Mark DB, Hague CJ, Min JK, Reynolds HR, Elghamaz A, Nair RG, Mavromatis K, Gosselin G, Banerjee S, Pejkov H, Lindsay S, Grantham JA, Williams DO, Stone GW, O'Brien SM, Hochman JS, Maron DJ; ISCHEMIA Research Group. Invasive vs Conservative Management of Patients With Chronic Total Occlusion: Results From the ISCHEMIA Trial. J Am Coll Cardiol. 2025 Apr 1;85(12):1335-1349. doi: 10.1016/j.jacc.2025.01.029. PMID 40139890
- [Derived] Maron DJ, Newman JD, Anthopolos R, Lu Y, Stevens S, Boden WE, Mavromatis K, Linefsky J, Nair RG, Bockeria O, Gosselin G, Perna GP, Demchenko E, Foo D, Shapiro MD, Champagne MA, Ballantyne C, McCullough P, Lopez-Sendon JL, Rockhold F, Harrell F, Rosenberg Y, Stone GW, Bangalore S, Reynolds HR, Spertus JA, Hochman JS; ISCHEMIA Research Group. Guideline-Directed Medical Therapy and Outcomes in the ISCHEMIA Trial. J Am Coll Cardiol. 2025 Apr 1;85(12):1317-1331. doi: 10.1016/j.jacc.2025.01.028. PMID 40139888
- [Derived] Slater J, Maron DJ, Jones PG, Bangalore S, Reynolds HR, Fu Z, Stone GW, Kirby R, Hochman JS, Spertus JA; ISCHEMIA Research Group. Evaluating the Appropriate Use Criteria for Coronary Revascularization in Stable Ischemic Heart Disease Using Randomized Data From the ISCHEMIA Trial. Circ Cardiovasc Qual Outcomes. 2025 Mar;18(3):e010849. doi: 10.1161/CIRCOUTCOMES.124.010849. Epub 2025 Feb 26. PMID 40008421
- [Derived] Hausvater A, Anthopolos R, Seltzer A, Spruill TM, Spertus JA, Peteiro J, Lopez-Sendon JL, Celutkiene J, Demchenko EA, Kedev S, Beleslin BD, Sidhu MS, Grodzinsky A, Fleg JL, Maron DJ, Hochman JS, Reynolds HR; CIAO-ISCHEMIA Research Group. Sex Differences in Psychosocial Factors and Angina in Patients With Chronic Coronary Disease. J Am Heart Assoc. 2025 Mar 4;14(5):e037909. doi: 10.1161/JAHA.124.037909. Epub 2025 Feb 25. PMID 39996455
- [Derived] Reynolds HR, Page CB, Shaw LJ, Berman DS, Chaitman BR, Picard MH, Kwong RY, Min JK, Leipsic J, Mancini GBJ, Budoff MJ, Hague CJ, Senior R, Szwed H, Bhargava B, Celutkiene J, Gadkari M, Bainey KR, Doerr R, Ramos RB, Ong P, Naik SR, Steg PG, Goetschalckx K, Chow BJW, Scherrer-Crosbie M, Phillips L, Mark DB, Spertus JA, Alexander KP, O'Brien SM, Boden WE, Bangalore S, Stone GW, Maron DJ, Hochman JS; ISCHEMIA Research Group. Relationship Between Severity of Ischemia and Coronary Artery Disease for Different Stress Test Modalities in the ISCHEMIA Trial. Circ Cardiovasc Interv. 2024 Dec;17(12):e013743. doi: 10.1161/CIRCINTERVENTIONS.123.013743. Epub 2024 Dec 17. PMID 39689188
- [Derived] Bangalore S, Rhodes G, Maron DJ, Anthopolos R, O'Brien SM, Jones PG, Mark DB, Reynolds HR, Spertus JA, Stone GW, White HD, Xu Y, Fremes SE, Hochman JS, Ischemia Research Group OBOT. Outcomes with revascularisation versus conservative management of participants with 3-vessel coronary artery disease in the ISCHEMIA trial. EuroIntervention. 2024 Oct 21;20(20):e1276-e1287. doi: 10.4244/EIJ-D-24-00240. PMID 39432255
- [Derived] Ikemura N, Spertus JA, Nguyen D, Fu Z, Jones PG, Reynolds HR, Bangalore S, Bhargava B, Senior R, Elghamaz A, Goodman SG, Lopes RD, Pracon R, Lopez-Sendon J, Maggioni AP, Kohsaka S, Roth GA, White HD, Mavromatis K, Boden WE, Rodriguez F, Hochman JS, Maron DJ; ISCHEMIA Research Group. International Variation in Health Status Benefits in Patients Undergoing Initial Invasive Versus Conservative Management for Chronic Coronary Disease: Insights From the ISCHEMIA Trial. Circ Cardiovasc Qual Outcomes. 2024 Oct;17(10):e010534. doi: 10.1161/CIRCOUTCOMES.123.010534. Epub 2024 Sep 20. PMID 39301726
- [Derived] Jorda A, Pecho T, Horvath LC, Nishani E, Bull LE, Bergmann F, Nitsche C, Zeitlinger M, Jilma B, Gelbenegger G. Association of Electrocardiogram Findings With Clinical Outcomes in Patients With Chronic Coronary Syndrome: An Analysis of the ISCHEMIA Trials. Am J Med. 2025 Jan;138(1):61-69.e3. doi: 10.1016/j.amjmed.2024.09.007. Epub 2024 Sep 14. PMID 39284482
- [Derived] Fleg JL, Huang Z, Reynolds HR, Shaw LJ, Chaitman BR, O'Brien SM, Berstein L, Peteiro J, Smanio PEP, Wander GS, Berger JS, Berman DS, Picard MH, Kwong RY, Min JK, Phillips LM, Bangalore S, Maron DJ, Hochman JS; ISCHEMIA Research Group. Ischemia Severity, Coronary Artery Disease Extent, and Exercise Capacity in ISCHEMIA. Circulation. 2024 Jul 9;150(2):165-167. doi: 10.1161/CIRCULATIONAHA.123.066980. Epub 2024 Jul 8. No abstract available. PMID 38976607
- [Derived] Jorda A, Hengstenberg C, Lang IM, Kautzky-Willer A, Harreiter J, Zeitlinger M, Jilma B, Gelbenegger G. Association of prediabetes with clinical outcomes in patients with chronic coronary syndrome: a post hoc analysis of the ISCHEMIA and ISCHEMIA-CKD trials. Cardiovasc Diabetol. 2024 May 20;23(1):176. doi: 10.1186/s12933-024-02232-z. PMID 38769562
- [Derived] Pracon R, Spertus JA, Broderick S, Bangalore S, Rockhold FW, Ruzyllo W, Demchenko E, Nageh T, Grossman GB, Mavromatis K, Manjunath CN, Smanio PEP, Stone GW, Mancini GBJ, Boden WE, Newman JD, Reynolds HR, Hochman JS, Maron DJ; ISCHEMIA Research Group. Factors Associated With Coronary Angiography Performed Within 6 Months of Randomization to the Conservative Strategy in the ISCHEMIA Trial. Circ Cardiovasc Interv. 2024 Jun;17(6):e013435. doi: 10.1161/CIRCINTERVENTIONS.123.013435. Epub 2024 Apr 17. PMID 38629312
- [Derived] Arnold SV, Jones PG, Maron DJ, Cohen DJ, Mark DB, Reynolds HR, Bangalore S, Chen J, Newman JD, Harrington RA, Stone GW, Hochman JS, Spertus JA; ISCHEMIA Research Group. Variation in Health Status With Invasive vs Conservative Management of Chronic Coronary Disease. J Am Coll Cardiol. 2024 Apr 16;83(15):1353-1366. doi: 10.1016/j.jacc.2024.02.019. PMID 38599711
- [Derived] Reynolds HR, Cyr DD, Merz CNB, Shaw LJ, Chaitman BR, Boden WE, Alexander KP, Rosenberg YD, Bangalore S, Stone GW, Held C, Spertus J, Goetschalckx K, Bockeria O, Newman JD, Berger JS, Elghamaz A, Lopes RD, Min JK, Berman DS, Picard MH, Kwong RY, Harrington RA, Thomas B, O'Brien SM, Maron DJ, Hochman JS; ISCHEMIA Research Group *. Sex Differences in Revascularization, Treatment Goals, and Outcomes of Patients With Chronic Coronary Disease: Insights From the ISCHEMIA Trial. J Am Heart Assoc. 2024 Mar 5;13(5):e029850. doi: 10.1161/JAHA.122.029850. Epub 2024 Feb 27. PMID 38410945
- [Derived] Mavromatis K, Jones PG, Ali ZA, Stone GW, Rhodes GM, Bangalore S, O'Brien S, Genereux P, Horst J, Dressler O, Goodman S, Alexander K, Mathew A, Chen J, Bhargava B, Uxa A, Boden WE, Mark DB, Reynolds HR, Maron DJ, Hochman JS, Spertus JA; ISCHEMIA Research Group. Complete Revascularization and Angina-Related Health Status in the ISCHEMIA Trial. J Am Coll Cardiol. 2023 Jul 25;82(4):295-313. doi: 10.1016/j.jacc.2023.05.025. PMID 37468185
- [Derived] Stone GW, Ali ZA, O'Brien SM, Rhodes G, Genereux P, Bangalore S, Mavromatis K, Horst J, Dressler O, Poh KK, Nath RK, Moorthy N, Witkowski A, Dwivedi SK, Bockeria O, Chen J, Smanio PEP, Picard MH, Chaitman BR, Berman DS, Shaw LJ, Boden WE, White HD, Fremes SE, Rosenberg Y, Reynolds HR, Spertus JA, Hochman JS, Maron DJ; ISCHEMIA Research Group. Impact of Complete Revascularization in the ISCHEMIA Trial. J Am Coll Cardiol. 2023 Sep 19;82(12):1175-1188. doi: 10.1016/j.jacc.2023.06.015. Epub 2023 Jul 17. PMID 37462593
- [Derived] Nguyen DD, Spertus JA, Alexander KP, Newman JD, Dodson JA, Jones PG, Stevens SR, O'Brien SM, Gamma R, Perna GP, Garg P, Vitola JV, Chow BJW, Vertes A, White HD, Smanio PEP, Senior R, Held C, Li J, Boden WE, Mark DB, Reynolds HR, Bangalore S, Chan PS, Stone GW, Arnold SV, Maron DJ, Hochman JS; ISCHEMIA Research Group. Health Status and Clinical Outcomes in Older Adults With Chronic Coronary Disease: The ISCHEMIA Trial. J Am Coll Cardiol. 2023 May 2;81(17):1697-1709. doi: 10.1016/j.jacc.2023.02.048. PMID 37100486
- [Derived] Gala ABE, Curzen N. Is There Still a Place for Revascularisation in the Management of Stable Coronary Artery Disease Following the ISCHEMIA Trial? Heart Int. 2020 Aug 8;14(1):13-15. doi: 10.17925/HI.2020.14.1.13. eCollection 2020. PMID 36277662
- [Derived] Reynolds HR, Diaz A, Cyr DD, Shaw LJ, Mancini GBJ, Leipsic J, Budoff MJ, Min JK, Hague CJ, Berman DS, Chaitman BR, Picard MH, Hayes SW, Scherrer-Crosbie M, Kwong RY, Lopes RD, Senior R, Dwivedi SK, Miller TD, Chow BJW, de Silva R, Stone GW, Boden WE, Bangalore S, O'Brien SM, Hochman JS, Maron DJ; ISCHEMIA Research Group. Ischemia With Nonobstructive Coronary Arteries: Insights From the ISCHEMIA Trial. JACC Cardiovasc Imaging. 2023 Jan;16(1):63-74. doi: 10.1016/j.jcmg.2022.06.015. Epub 2022 Sep 14. PMID 36115814
- [Derived] Garcia RA, Spertus JA, Benton MC, Jones PG, Mark DB, Newman JD, Bangalore S, Boden WE, Stone GW, Reynolds HR, Hochman JS, Maron DJ; ISCHEMIA Research Group. Association of Medication Adherence With Health Outcomes in the ISCHEMIA Trial. J Am Coll Cardiol. 2022 Aug 23;80(8):755-765. doi: 10.1016/j.jacc.2022.05.045. PMID 35981820
- [Derived] Bangalore S, Spertus JA, Stevens SR, Jones PG, Mancini GBJ, Leipsic J, Reynolds HR, Budoff MJ, Hague CJ, Min JK, Boden WE, O'Brien SM, Harrington RA, Berger JS, Senior R, Peteiro J, Pandit N, Bershtein L, de Belder MA, Szwed H, Doerr R, Monti L, Alfakih K, Hochman JS, Maron DJ; ISCHEMIA Research Group. Outcomes With Intermediate Left Main Disease: Analysis From the ISCHEMIA Trial. Circ Cardiovasc Interv. 2022 Apr;15(4):e010925. doi: 10.1161/CIRCINTERVENTIONS.121.010925. Epub 2022 Apr 12. PMID 35411785
- [Derived] Mark DB, Spertus JA, Bigelow R, Anderson S, Daniels MR, Anstrom KJ, Baloch KN, Cohen DJ, Held C, Goodman SG, Bangalore S, Cyr D, Reynolds HR, Alexander KP, Rosenberg Y, Stone GW, Maron DJ, Hochman JS; ISCHEMIA Research Group. Comprehensive Quality-of-Life Outcomes With Invasive Versus Conservative Management of Chronic Coronary Disease in ISCHEMIA. Circulation. 2022 Apr 26;145(17):1294-1307. doi: 10.1161/CIRCULATIONAHA.121.057363. Epub 2022 Mar 9. PMID 35259918
- [Derived] Senior R, Reynolds HR, Min JK, Berman DS, Picard MH, Chaitman BR, Shaw LJ, Page CB, Govindan SC, Lopez-Sendon J, Peteiro J, Wander GS, Drozdz J, Marin-Neto J, Selvanayagam JB, Newman JD, Thuaire C, Christopher J, Jang JJ, Kwong RY, Bangalore S, Stone GW, O'Brien SM, Boden WE, Maron DJ, Hochman JS; ISCHEMIA Research Group. Predictors of Left Main Coronary Artery Disease in the ISCHEMIA Trial. J Am Coll Cardiol. 2022 Feb 22;79(7):651-661. doi: 10.1016/j.jacc.2021.11.052. PMID 35177194
- [Derived] Newman JD, Anthopolos R, Mancini GBJ, Bangalore S, Reynolds HR, Kunichoff DF, Senior R, Peteiro J, Bhargava B, Garg P, Escobedo J, Doerr R, Mazurek T, Gonzalez-Juanatey J, Gajos G, Briguori C, Cheng H, Vertes A, Mahajan S, Guzman LA, Keltai M, Maggioni AP, Stone GW, Berger JS, Rosenberg YD, Boden WE, Chaitman BR, Fleg JL, Hochman JS, Maron DJ. Outcomes of Participants With Diabetes in the ISCHEMIA Trials. Circulation. 2021 Oct 26;144(17):1380-1395. doi: 10.1161/CIRCULATIONAHA.121.054439. Epub 2021 Sep 15. PMID 34521217
- [Derived] Lopez-Sendon JL, Cyr DD, Mark DB, Bangalore S, Huang Z, White HD, Alexander KP, Li J, Nair RG, Demkow M, Peteiro J, Wander GS, Demchenko EA, Gamma R, Gadkari M, Poh KK, Nageh T, Stone PH, Keltai M, Sidhu M, Newman JD, Boden WE, Reynolds HR, Chaitman BR, Hochman JS, Maron DJ, O'Brien SM. Effects of initial invasive vs. initial conservative treatment strategies on recurrent and total cardiovascular events in the ISCHEMIA trial. Eur Heart J. 2022 Jan 13;43(2):148-149. doi: 10.1093/eurheartj/ehab509. PMID 34514494
- [Derived] Reynolds HR, Shaw LJ, Min JK, Page CB, Berman DS, Chaitman BR, Picard MH, Kwong RY, O'Brien SM, Huang Z, Mark DB, Nath RK, Dwivedi SK, Smanio PEP, Stone PH, Held C, Keltai M, Bangalore S, Newman JD, Spertus JA, Stone GW, Maron DJ, Hochman JS. Outcomes in the ISCHEMIA Trial Based on Coronary Artery Disease and Ischemia Severity. Circulation. 2021 Sep 28;144(13):1024-1038. doi: 10.1161/CIRCULATIONAHA.120.049755. Epub 2021 Sep 9. PMID 34496632
- [Derived] White HD, O'Brien SM, Alexander KP, Boden WE, Bangalore S, Li J, Manjunath CN, Lopez-Sendon JL, Peteiro J, Gosselin G, Berger JS, Maggioni AP, Reynolds HR, Hochman JS, Maron DJ. Comparison of Days Alive Out of Hospital With Initial Invasive vs Conservative Management: A Prespecified Analysis of the ISCHEMIA Trial. JAMA Cardiol. 2021 Sep 1;6(9):1023-1031. doi: 10.1001/jamacardio.2021.1651. PMID 33938917
- [Derived] Chaitman BR, Alexander KP, Cyr DD, Berger JS, Reynolds HR, Bangalore S, Boden WE, Lopes RD, Demkow M, Piero Perna G, Riezebos RK, McFalls EO, Banerjee S, Bagai A, Gosselin G, O'Brien SM, Rockhold FW, Waters DD, Thygesen KA, Stone GW, White HD, Maron DJ, Hochman JS; ISCHEMIA Research Group. Myocardial Infarction in the ISCHEMIA Trial: Impact of Different Definitions on Incidence, Prognosis, and Treatment Comparisons. Circulation. 2021 Feb 23;143(8):790-804. doi: 10.1161/CIRCULATIONAHA.120.047987. Epub 2020 Dec 3. PMID 33267610
- [Derived] Lopes RD, Alexander KP, Stevens SR, Reynolds HR, Stone GW, Pina IL, Rockhold FW, Elghamaz A, Lopez-Sendon JL, Farsky PS, Chernyavskiy AM, Diaz A, Phaneuf D, De Belder MA, Ma YT, Guzman LA, Khouri M, Sionis A, Hausenloy DJ, Doerr R, Selvanayagam JB, Maggioni AP, Hochman JS, Maron DJ. Initial Invasive Versus Conservative Management of Stable Ischemic Heart Disease in Patients With a History of Heart Failure or Left Ventricular Dysfunction: Insights From the ISCHEMIA Trial. Circulation. 2020 Nov 3;142(18):1725-1735. doi: 10.1161/CIRCULATIONAHA.120.050304. Epub 2020 Aug 29. PMID 32862662
- [Derived] Maron DJ, Hochman JS, Reynolds HR, Bangalore S, O'Brien SM, Boden WE, Chaitman BR, Senior R, Lopez-Sendon J, Alexander KP, Lopes RD, Shaw LJ, Berger JS, Newman JD, Sidhu MS, Goodman SG, Ruzyllo W, Gosselin G, Maggioni AP, White HD, Bhargava B, Min JK, Mancini GBJ, Berman DS, Picard MH, Kwong RY, Ali ZA, Mark DB, Spertus JA, Krishnan MN, Elghamaz A, Moorthy N, Hueb WA, Demkow M, Mavromatis K, Bockeria O, Peteiro J, Miller TD, Szwed H, Doerr R, Keltai M, Selvanayagam JB, Steg PG, Held C, Kohsaka S, Mavromichalis S, Kirby R, Jeffries NO, Harrell FE Jr, Rockhold FW, Broderick S, Ferguson TB Jr, Williams DO, Harrington RA, Stone GW, Rosenberg Y; ISCHEMIA Research Group. Initial Invasive or Conservative Strategy for Stable Coronary Disease. N Engl J Med. 2020 Apr 9;382(15):1395-1407. doi: 10.1056/NEJMoa1915922. Epub 2020 Mar 30. PMID 32227755
- [Derived] Spertus JA, Jones PG, Maron DJ, O'Brien SM, Reynolds HR, Rosenberg Y, Stone GW, Harrell FE Jr, Boden WE, Weintraub WS, Baloch K, Mavromatis K, Diaz A, Gosselin G, Newman JD, Mavromichalis S, Alexander KP, Cohen DJ, Bangalore S, Hochman JS, Mark DB; ISCHEMIA Research Group. Health-Status Outcomes with Invasive or Conservative Care in Coronary Disease. N Engl J Med. 2020 Apr 9;382(15):1408-1419. doi: 10.1056/NEJMoa1916370. Epub 2020 Mar 30. PMID 32227753
- [Derived] Reynolds HR, Shaw LJ, Min JK, Spertus JA, Chaitman BR, Berman DS, Picard MH, Kwong RY, Bairey-Merz CN, Cyr DD, Lopes RD, Lopez-Sendon JL, Held C, Szwed H, Senior R, Gosselin G, Nair RG, Elghamaz A, Bockeria O, Chen J, Chernyavskiy AM, Bhargava B, Newman JD, Hinic SB, Jaroch J, Hoye A, Berger J, Boden WE, O'Brien SM, Maron DJ, Hochman JS; ISCHEMIA Research Group. Association of Sex With Severity of Coronary Artery Disease, Ischemia, and Symptom Burden in Patients With Moderate or Severe Ischemia: Secondary Analysis of the ISCHEMIA Randomized Clinical Trial. JAMA Cardiol. 2020 Jul 1;5(7):773-786. doi: 10.1001/jamacardio.2020.0822. PMID 32227128
- [Derived] Azevedo DFC, Lima EG, Ribeiro MOL, Linhares Filho JPP, Serrano Junior CV. Critical analysis of the classic indications for myocardial revascularization. Rev Assoc Med Bras (1992). 2019 Mar;65(3):319-325. doi: 10.1590/1806-9282.65.3.319. Epub 2019 Apr 11. PMID 30994826
- [Derived] Shaw LJ, Xie JX, Phillips LM, Goyal A, Reynolds HR, Berman DS, Picard MH, Bhargava B, Devlin G, Chaitman BR. Optimising diagnostic accuracy with the exercise ECG: opportunities for women and men with stable ischaemic heart disease. Heart Asia. 2016 Jun 1;8(2):1-7. doi: 10.1136/heartasia-2016-010736. eCollection 2016. PMID 27326241
- [Derived] Kataoka A, Scherrer-Crosbie M, Senior R, Gosselin G, Phaneuf D, Guzman G, Perna G, Lara A, Kedev S, Mortara A, El-Hajjar M, Shaw LJ, Reynolds HR, Picard MH. The value of core lab stress echocardiography interpretations: observations from the ISCHEMIA Trial. Cardiovasc Ultrasound. 2015 Dec 18;13:47. doi: 10.1186/s12947-015-0043-2. PMID 26683627
- [Derived] Stone GW, Hochman JS, Williams DO, Boden WE, Ferguson TB Jr, Harrington RA, Maron DJ. Medical Therapy With Versus Without Revascularization in Stable Patients With Moderate and Severe Ischemia: The Case for Community Equipoise. J Am Coll Cardiol. 2016 Jan 5;67(1):81-99. doi: 10.1016/j.jacc.2015.09.056. Epub 2015 Nov 23. PMID 26616030
- [Derived] Wasilewski J, Polonski L, Lekston A, Osadnik T, Regula R, Bujak K, Kurek A. Who is eligible for randomized trials? A comparison between the exclusion criteria defined by the ISCHEMIA trial and 3102 real-world patients with stable coronary artery disease undergoing stent implantation in a single cardiology center. Trials. 2015 Sep 15;16:411. doi: 10.1186/s13063-015-0934-4. PMID 26373291
- See also: Main Website for ISCHEMIA Trial — http://www.ischemiatrial.org/
- See also: Angioplasty — http://www.nlm.nih.gov/medlineplus/angioplasty.html
- See also: Coronary Artery Bypass Surgery — http://www.nlm.nih.gov/medlineplus/coronaryarterybypasssurgery.html
- See also: Coronary Artery Disease — http://www.nlm.nih.gov/medlineplus/coronaryarterydisease.html
- See also: Heart Diseases — http://www.nlm.nih.gov/medlineplus/heartdiseases.html
- See also: ISCHEMIA Trial Update — https://doi.org/10.1016/j.ahj.2019.09.001

RESULTS

PARTICIPANT FLOW:
Groups:
- Invasive Strategy (INV): Routine invasive strategy with cardiac catheterization followed by revascularization plus optimal medical therapy.
  Cardiac catheterization: Narrowed blood vessels can be opened without surgery using stents or bypassed with surgery. To determine the best approach, the doctor must assess the severity of blood vessel narrowings. This procedure is known as cardiac catheterization.
  Coronary artery bypass graft surgery: Artery narrowing is bypassed during surgery with a healthy artery or vein from another part of the body. This is known as coronary artery bypass grafting, or CABG (said, "cabbage"). The surgery creates new routes around narrowed and blocked heart arteries, allowing more blood flow to the heart.
  Percutaneous coronary intervention: done as part of the cardiac catheterization procedure. A small, hollow, mesh tube (stent) is inserted into the narrowed part of the artery. The stent pushes the plaque against the artery wall, and opens the vessel to allow better blood flow.
Period: Overall Study
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Started | 2588 | 2591
Completed | 2524 | 2543
Not Completed | 64 | 48
Not completed — Withdrawal by Subject | 28 | 22
Not completed — Lost to Follow-up | 36 | 26

BASELINE CHARACTERISTICS:
Groups:
- Invasive Strategy (INV): Invasive Strategy (INV)
- Conservative Strategy: Conservative Strategy
- Total: Total of all reporting groups
Arm/Group | Invasive Strategy (INV) | Conservative Strategy | Total
Number analyzed (Participants) | 2588 | 2591 | 5179
Age, Continuous [Mean (Full Range); unit: years] | 64 [58 to 70] | 64 [58 to 70] | 64 [58 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 606 | 562 | 1168
  Male | 1982 | 2029 | 4011
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 372 | 391 | 763
  Not Hispanic or Latino | 2030 | 2022 | 4052
  Unknown or Not Reported | 186 | 178 | 364
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 5 | 13
  Asian | 747 | 738 | 1485
  Native Hawaiian or Other Pacific Islander | 5 | 7 | 12
  Black or African American | 96 | 108 | 204
  White | 1706 | 1697 | 3403
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 19 | 31 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  Africa | 8 | 5 | 13
  Asia | 791 | 786 | 1577
  Europe | 853 | 865 | 1718
  Latin America | 239 | 239 | 478
  Middle East | 10 | 10 | 20
  North America | 648 | 652 | 1300
  Pacifica | 39 | 34 | 73

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Outcome: Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, Heart Failure, or Resuscitated Cardiac Arrest
Time Frame: 3.2 year follow-up (median)
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Participants | 318 | 352

2. Primary Outcome: Cumulative Event Rate of Primary Composite Outcome (Death From Cardiovascular Causes, Myocardial Infarction, or Hospitalization for Unstable Angina, Heart Failure, or Resuscitated Cardiac Arrest)
Description: This measure represents the estimated cumulative probability of experiencing the primary endpoint within the indicated timeframe in each treatment group. The interpretation of the measure is similar to Kaplan-Meier event rates. Estimates are expressed as percentages ranging from 0% (endpoint is certain not to occur) to 100% (endpoint is certain to occur).
Time Frame: 5 years
Measure: Number; unit: cumulative event rate - %
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
cumulative event rate - %
  At 6 months | 5.3 | 3.4
  At 1 year | 7.0 | 5.4
  At 2 years | 9.0 | 9.5
  At 3 years | 11.3 | 12.7
  At 4 years | 13.3 | 15.5
  At 5 years | 16.4 | 18.2

3. Primary Outcome: Number of Participants That Experienced Death From Cardiovascular Causes or Myocardial Infarction
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Participants | 276 | 314

4. Primary Outcome: Cumulative Event Rate of Death From Cardiovascular Causes or Myocardial Infarction
Description: This measure represents the estimated cumulative probability of experiencing Death from cardiovascular causes or myocardial infarction within the indicated timeframe in each treatment group. The interpretation of the measure is similar to Kaplan-Meier event rates. Estimates are expressed as percentages ranging from 0% (endpoint is certain not to occur) to 100% (endpoint is certain to occur).
Time Frame: 5 years
Measure: Number; unit: Cumulative event rate -- %
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Cumulative event rate -- %
  At 6 months | 4.8 | 2.9
  At 1 year | 6.2 | 4.6
  At 2 years | 7.9 | 8.2
  At 3 years | 9.7 | 11.0
  At 4 years | 11.7 | 13.9
  At 5 years | 14.2 | 16.5

5. Primary Outcome: Number of Participants That Experienced Death From Any Cause
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Participants | 145 | 144

6. Primary Outcome: Cumulative Event Rate of Death From Any Cause
Time Frame: 5 years
Measure: Number; unit: Cumulative event rate -- %
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Cumulative event rate -- %
  At 6 months | 0.8 | 0.4
  At 1 year | 1.7 | 1.0
  At 2 years | 2.8 | 2.9
  At 3 years | 4.3 | 4.3
  At 4 years | 6.5 | 6.4
  At 5 years | 9.0 | 8.3

7. Primary Outcome: Number of Participants That Experienced Myocardial Infarction
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Participants | 210 | 233

8. Primary Outcome: Cumulative Event Rate of Myocardial Infarction
Time Frame: 5 years
Measure: Number; unit: Cumulative event rate -- %
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
Number analyzed (Participants) | 2588 | 2591
Cumulative event rate -- %
  At 6 months | 4.3 | 2.6
  At 1 year | 5.3 | 3.8
  At 2 years | 6.3 | 6.5
  At 3 years | 7.7 | 8.5
  At 4 years | 8.9 | 10.1
  At 5 years | 10.3 | 11.9

9. Primary Outcome: Estimated Difference in Cumulative Event Rate ( %) of Primary Composite Outcome: Invasive Minus Conservative
Description: The primary composite outcome includes death from cardiovascular causes, myocardial infarction, or hospitalization for unstable angina, heart failure, or resuscitated cardiac arrest.
Time Frame: 5 years
Population: Invasive = 2588; Conservative = 2591
Measure: Number (95% Confidence Interval); unit: cumulative event rate - %
Groups:
- Between Invasive and Conservative Strategy Arms: Invasive vs. Conservative
Arm/Group | Between Invasive and Conservative Strategy Arms
Number analyzed (Participants) | 5179
cumulative event rate - %
  At 6 months | 1.9 [0.8 to 3.0]
  At 1 year | 1.5 [0.2 to 2.9]
  At 2 years | -0.5 [-2.1 to 1.1]
  At 3 years | -1.3 [-3.2 to 0.6]
  At 4 years | -2.2 [-4.4 to 0]
  At 5 years | -1.8 [-4.7 to 1.0]

10. Primary Outcome: Estimated Difference in Cumulative Event Rate of Death From Cardiovascular Causes: Invasive Minus Conservative or Myocardial Infarction Between Invasive and Conservative Strategies
Time Frame: 5 years
Population: Invasive = 2588; Conservative = 2591
Measure: Number (95% Confidence Interval); unit: cumulative event rate - %
Arm/Group | Between Invasive and Conservative Strategy Arms
Number analyzed (Participants) | 5179
cumulative event rate - %
  At 6 months | 1.9 [0.9 to 3.0]
  At 1 year | 1.6 [0.4 to 2.8]
  At 2 years | -0.3 [-1.8 to 1.2]
  At 3 years | -1.3 [-3.1 to 0.5]
  At 4 years | -2.2 [-4.4 to -0.1]
  At 5 years | -2.3 [-5.0 to 0.4]

11. Primary Outcome: Estimated Difference in Cumulative Event Rate of Death From Any Cause: Invasive Minus Conservative
Time Frame: 5 years
Population: Invasive = 2588; Conservative = 2591
Measure: Number (95% Confidence Interval); unit: cumulative event rate - %
Arm/Group | Between Invasive and Conservative Strategy Arms
Number analyzed (Participants) | 5179
cumulative event rate - %
  At 6 months | 0.4 [0 to 0.8]
  At 1 year | 0.7 [0 to 1.3]
  At 2 years | -0.1 [-1.0 to 0.9]
  At 3 years | 0 [-1.2 to 1.2]
  At 4 years | 0.1 [-1.5 to 1.8]
  At 5 years | 0.7 [-1.6 to 3.1]

12. Primary Outcome: Estimated Difference in Cumulative Event Rate of Myocardial Infarction: Invasive Minus Conservative
Time Frame: 5 years
Population: Invasive = 2588; Conservative = 2591
Measure: Number (95% Confidence Interval); unit: cumulative event rate - %
Arm/Group | Between Invasive and Conservative Strategy Arms
Number analyzed (Participants) | 5179
cumulative event rate - %
  At 6 months | 1.8 [0.8 to 2.8]
  At 1 year | 1.5 [0.3 to 2.6]
  At 2 years | -0.1 [-1.5 to 1.2]
  At 3 years | -0.7 [-2.3 to 0.8]
  At 4 years | -1.2 [-3.0 to 0.6]
  At 5 years | -1.6 [-3.9 to 0.7]

ADVERSE EVENTS:
Time Frame: 5 years
Description: SAEs were collected as part of the Primary Composite Outcome
Arm/Group | Invasive Strategy (INV) | Conservative Strategy
All-Cause Mortality (participants affected / at risk) | 145/2588 | 144/2591
Serious Adverse Events (participants affected / at risk) | 318/2588 | 352/2591
Other Adverse Events (participants affected / at risk) | 0/2588 | 0/2591
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Invasive Strategy (INV) (N=2588) | Conservative Strategy (N=2591)
Cardiovascular Death (Cardiac disorders) | 92 (92) | 111 (111)
Procedural Myocardial Infarction (Cardiac disorders) | 70 (70) | 24 (24)
Non-procedural Myocardial Infarction (Cardiac disorders) | 130 (130) | 196 (196)
Hospitalization for Unstable Angina (Cardiac disorders) | 16 (16) | 32 (32)
Hospitalization for Heart Failure (Cardiac disorders) | 51 (51) | 25 (25)
Resuscitated Cardiac Arrest (Cardiac disorders) | 5 (5) | 5 (5)
Stroke (Cardiac disorders) | 45 (45) | 38 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Study Protocol v.1.0 (2012-01-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT01471522/Prot_000.pdf
  • Study Protocol: Study Protocol v.2.0 (2014-01-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT01471522/Prot_001.pdf
  • Study Protocol: Protocol Addendum (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT01471522/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT01471522/SAP_003.pdf